CLINICAL TRIAL: NCT01440582
Title: Phase I/Ib Trial of the Efficacy and Safety of Combination Therapy of Lenalidomide/Bortezomib/Dexamethasone and Panobinostat in Transplant Eligible Patients With Newly Diagnosed Multiple Myeloma (MM)
Brief Title: Combination Therapy of Lenalidomide/Bortezomib/Dexamethasone and Panobinostat in Transplant Eligible New Diagnosed Multiple Myeloma (MM) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0192; NCI-2015-01566 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Myeloma
Keywords: Myeloma; Multiple Myeloma; MM; Newly diagnosed; Transplant eligible; Panobinostat; LBH589B; Bortezomib; Velcade; LDP-341; MLN341; PS-341; Lenalidomide; CC-5013; Revlimid; Dexamethasone; Decadron; Symptom questionnaire; Survey
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Panobinostat; Bortezomib; Lenalidomide; Dexamethasone; Calcium Dobesilate; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat + Bortezomib + Lenalidomide + Dexamethasone (Experimental): Induction Starting Doses: Lenalidomide 25 mg orally daily on days 1-14; Bortezomib 1.3 mg/m^2 intravenous (IV) daily on days 1, 4, 8 and 11; Dexamethasone 20 mg orally daily on days 1, 2, 4, 5, 8, 9, 11, 12 and Panobinostat orally 10 mg on days 1, 3, 5, 8, 10 and 12. Induction therapy consists of 21 day cycle in Part A and 28 day cycle in Part B.
  Symptom Questionnaire completed on day 1 of each cycle.
  Interventions: Drug: Panobinostat; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Behavioral: Symptom Questionnaire

INTERVENTIONS:
Drug: Panobinostat — Induction Therapy (Part A, 21-day cycles): 10 mg by mouth on Days 1, 3, 5, 8, 10, and 12 for 2 weeks with 1 week of rest at the end of each cycle.
  Induction Therapy (Part B, 28-day cycles): 10 mg by mouth on Days 1, 3, 5, 15, 17, and 19 of every cycle.
  Maintenance dose (Part A, 28-day cycles): Maximum tolerated dose (MTD) from Induction phase on Days 1, 3, 5, 8, 10, and 12 of each cycle.
  Maintenance dose (Part B, 28-day cycles): Maximum tolerated dose (MTD) from Induction phase on Days 1, 3, 5, 15, 17, 19 of each cycle.
  Other Names: LBH589B
Drug: Bortezomib — Induction Therapy (Part A, 21-day cycles): 1.3 mg/m^2 by vein daily on days 1, 4, 8 and 11 of Cycles 1 - 8.
  Induction Therapy (Part B, 28-day cycles): 1.3 mg/m^2 by vein daily on days 1, 8 and 15 of Cycles 1 - 8.
  Other Names: Velcade; LDP-341; MLN341; PS-341
Drug: Lenalidomide — Induction Therapy (Part A, 21-day cycles): 25 mg by mouth daily on days 1-14 of every cycle.
  Induction Therapy (Part B, 28-day cycles): 25 mg by mouth daily on days 1-21 of every cycle.
  Maintenance dose (Parts A and B, 28-day cycles): Last tolerated dose from Induction Phase on Days 1 - 21 of each cycle.
  Other Names: CC-5013; Revlimid
Drug: Dexamethasone — Induction Therapy (Part A, 21-day cycles): 20 mg by mouth daily on Days 1, 2, 4, 5, 8, 9, 11 and 12 of Cycles 1 - 8.
  Induction Therapy (Part B, 28-day cycles): 20 mg by mouth daily on Days 1, 2, 8, 9, 15 and 16 of Cycles 1-8.
  Maintenance dose (Parts A and B, 28-day cycles): Last tolerated dose from Induction Phase on Days 1, 8, 15, 21 of each cycle.
  Other Names: Decadron
Behavioral: Symptom Questionnaire — Completed on day 1 of each cycle.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the drug panobinostat that can be given in combination with the drugs Velcade (bortezomib), Revlimid (lenalidomide), and Decadron (dexamethasone) to patients with MM. The safety of this drug combination will also be studied.

Panobinostat is designed to cause chemical changes in different groups of proteins that are attached to DNA (the genetic material of cells), which may slow the growth of cancer cells or cause the cancer cells to die.

Bortezomib is designed to block a protein that causes cells to grow. This may cause cancer cells to die.

Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. This may slow the growth of cancer cells.

Dexamethasone is a corticosteroid that is similar to a natural hormone made by your body. Dexamethasone is often given to MM patients in combination with other chemotherapy to treat cancer.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of panobinostat based on when you join this study.

If you are enrolled in the first portion of Part A, up to 4 dose levels of panobinostat will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of panobinostat is found.

If you are enrolled in the second portion of Part A, you will receive panobinostat at the recommended dose from the first portion of Part A.

If you are enrolled in the first portion of Part B, up to 3 dose levels of panobinostat will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of panobinostat is found.

If you are enrolled in the second portion of Part B, you will receive panobinostat at the recommended dose from the first portion of Part B.

Study Drug Administration:

Induction Therapy (Part A):

In the Induction phase of therapy, each cycle is 21 days.

On Days 1, 4, 8, and 11 of Cycles 1-8, you will receive bortezomib either through a needle under your skin or by vein over 3-5 seconds. You will be watched by the study staff for 30 minutes after the infusion.

On Days 1-14 of every cycle, you will take lenalidomide by mouth 1 time each day. You should swallow the lenalidomide capsules whole with 1 cup (about 8 ounces) of water. Do not break, chew, or open the capsules.

You will take panobinostat by mouth 1 time a day with food on Days 1, 3, 5, 8, 10 and 12 for 2 weeks with 1 week of rest at the end of each cycle.

On Days 1, 2, 4, 5, 8, 9, 11, and 12 of Cycles 1-8, you will take dexamethasone by mouth 1 time a day. After 8 cycles, you may continue to take dexamethasone if the doctor thinks it is needed. Dexamethasone should be taken with food.

Induction Therapy (Part B):

In Part B, the induction phase of therapy is 28-day cycles.

On Days 1, 8, and 15 of Cycles 1-8, you will receive bortezomib either through a needle under your skin or by vein over 3-5 seconds. You will be watched by the study staff for 30 minutes after the infusion.

On Days 1-21 of every cycle, you will take lenalidomide by mouth 1 time each day. You should swallow the lenalidomide capsules whole with 1 cup (about 8 ounces) of water. Do not break, chew, or open the capsules.

You will take panobinostat by mouth 1 time a day with food on Days 1, 3, 5, 15, 17, 19 of every cycle.

On Days 1, 2, 8, 9, 15,16, Cycles 1-8, you will take dexamethasone by mouth 1 time a day. After 8 cycles, you may continue to take dexamethasone if the doctor thinks it is needed. Dexamethasone should be taken with food.

Maintenance Therapy (Parts A and B):

In the Maintenance phase of therapy, each cycle is 28 days.

You will take lenalidomide by mouth 1 time each day on Days 1-21 of each cycle.

You will take dexamethasone by mouth 1 time a day on Days 1, 8, 15, and 21 of each cycle.

In Part A, you will take panobinostat by mouth 1 time a day on Days 1, 3, 5, 8, 10, and 12 of each cycle. In Part B, you will take panobinostat by mouth 1 time a day on Days 1, 3, 5, 15, 17, 19 of each cycle.

Other Instructions:

You can take the study drugs anytime during the day but you should take them at the same time every day.

If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose). If you take more than the prescribed dose of lenalidomide, you should seek emergency medical care if needed and contact the study staff right away.

Your study drug doses may be lowered if you have side effects.

You will be given a drug diary for each cycle to write in to help keep track of your study drug doses. You should bring the drug diary and pill bottles to your study visit at the beginning of each new cycle.

The panobinostat capsule(s) should be swallowed with 1 cup of water. You should try to take the dose at around the same time each day. If you vomit after taking panobinostat, you should not take it again until your next scheduled dose. If you forget to take a dose in the morning, you can take it up to 12 hours later. If you miss a dose for more than 12 hours, you should wait until your next scheduled dose. Do not make up missed doses.

On Day 1 of every new study cycle and Cycle 1, Day 5, you should wait to take your panobinostat until you come to the clinic for study tests. Some of the Day 1 tests need to be performed before dosing.

You need to follow all panobinostat dosing instructions as written. Do not miss any panobinostat capsules. You will be asked to return all unused study drug in the bottles provided, along with empty bottles, on Day 1 of every cycle, starting with Cycle 2. Capsules should not be transferred between bottles at any time. Please do not allow anyone else to handle or touch the study drug.

You can stop anytime after Cycle 4 of Induction to have a stem cell transplant. If you decide with your doctor to delay the transplant, you will still be recommended to have your stem cells collected. You will continue with Induction therapy until you have had 4-8 cycles. After that, you will receive Maintenance therapy.

You will be given other drugs to help prevent side effects. The study staff will tell you about these drugs, how they will be given, and the possible risks.

Study Visits (Part A):

On Day 1 of each cycle:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 5 tablespoons) will be drawn for routine tests and biomarker testing.
* Blood (about 1 teaspoon) and/or urine will be collected to check the status of the disease. If urine is collected, you will collect the urine over 24 hours. This urine or blood will also be used for a pregnancy test if you are able to become pregnant.
* You will complete the symptom questionnaire.
* You will be asked about any symptoms you may have had and any drugs you may be taking.
* If the doctor thinks it is needed, you will have bone x-rays, an MRI and/or a CT scan to check the status of the disease.

On Days 1 and 5 of Cycle 1, you will have 3 ECGs before the study drug dose and 3 ECGs after the dose.

On Day 1 of Cycles 2-8, you will have 3 ECGs.

On Days 4, 8, and 11 of Cycles 1-8:

°Blood (about 4 tablespoons) will be drawn for routine tests.

At the end of Cycle 8 (or if you are going to have a stem cell transplant, at the end of Cycle 4):

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any symptoms you may have had and any other drugs you may be taking.
* Blood (about 2 tablespoons) will be collected for routine tests.
* Blood (about 1 teaspoon) and/or urine will be collected to check the status of the disease. If urine is collected, you will be asked to collect your urine over 24 hours.
* You will have bone x-rays to check the status of the disease.
* If the disease completely responds to the study drugs, you will have a bone marrow aspiration and/or biopsy to confirm the response.

On Day 1 of Maintenance Therapy, or Cycles 9 and beyond (if you choose to delay stem cell transplant) :

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any symptoms you may have had and any other drugs you may be taking.
* You will complete the symptom questionnaire.
* Blood (about 4 tablespoons) will be drawn for routine tests and biomarker testing.
* Blood (about 1 teaspoon) and/or urine will be collected to check the status of the disease. If urine is collected, you will collect the urine for 24 hours. This urine or blood will also be used for a pregnancy test if you are able to become pregnant.
* If the doctor thinks it is needed, you will have bone x-rays, an MRI and/or a CT scan to check the status of the disease.

Study Visits (Part B):

On Days 8 and 15 of Cycle 1, blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 2 and beyond:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any symptoms you may have had and any other drugs you may be taking.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* You will have 3 ECGs.

Pregnancy Tests (Parts A and B):

During induction therapy, if you are a woman who is able to become pregnant and you have regular or no periods, you will have a blood (about 1 tablespoon) or urine pregnancy test weekly for the first 21 days and then every 21 days while on therapy (including breaks in therapy). If you are a woman who is able to become pregnant and your cycles are irregular, you will have a blood (about 1 tablespoon) or urine pregnancy test weekly for the first 21 days during then every 11-14 days while on therapy (including breaks in therapy).

During maintenance therapy, if you are a woman who is able to become pregnant and have regular or no menstruation, you must have a pregnancy test every 28 days while on therapy (including breaks in therapy). If you are a woman who is able to become pregnant and your cycles are irregular, you will have a blood (about 1 tablespoon) or urine pregnancy test every 14 days (+/-1 day) and every 28 days.

Length of Treatment:

You may receive induction therapy for up to 8 cycles, followed by maintenance therapy for an additional 2 years. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment and follow-up visits.

End-of-Treatment Visit:

Within 30 days after your last dose of study drugs:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any symptoms you may be experiencing.
* Blood (about 4 tablespoon) and urine will be collected for routine tests.
* Blood (about 1 teaspoon) and/or urine will be collected to check the status of the disease. If urine is collected, you will collect the urine for 24 hours.
* If the disease completely responds to the study drugs, you will have a bone marrow aspiration and/or biopsy to confirm the response.
* If the doctor thinks it is needed, you will have an MRI and/or a CT scan to check the status of the disease.
* If you are able to become pregnant, you will have a urine or blood (about 1 tablespoon) pregnancy test.

Follow-Up:

Every 3 months (+/-1 month) for the first 2 years after the stem cell transplant and then every 6 months (+/- 2 months) for Years 3 and 4, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 4 tablespoons) and urine will be collected for routine tests.
* If the doctor thinks it is needed, you will also have an MRI and/or a CT scan, x-rays, and/or a bone marrow aspiration and biopsy.

Every 6 months during the first 2 years after you are finished with maintenance therapy, you will be asked how you are doing. This will be done at the clinic or by a phone call from the study staff. If you are called, the calls should take 5-10 minutes.

If the disease gets worse, you will no longer have follow-up.

This is an investigational study. Panobinostat is not FDA approved or commercially available. It is currently being used for research purposes only. Bortezomib is FDA approved and commercially available for the treatment of MM. Lenalidomide is FDA approved and commercially available for the treatment of certain types of myelodysplastic syndrome and for MM. The use of this drug combination to treat MM is investigational.

Up to 54 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Clonal bone marrow plasma cells >/=10% or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following myeloma defining events: Myeloma defining events: Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically: Hypercalcaemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11 mg/dL) Renal insufficiency: creatinine clearance <40 mL per min† or serum creatinine >177 μmol/L (>2 mg/dL)Anaemia: haemoglobin value of >20 g/L below the lower limit of normal, or a haemoglobin value <100 g/L Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET-CT Any one or more of the following biomarkers of malignancy: Clonal bone marrow plasma cell percentage ≥60% Involved:uninvolved serum free light chain ratio§ ≥100>1 focal lesions on MRI studies.
2. Continue of Inclusion Criteria 1: If bone marrow has less than 10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement. Patient must not have been previously treated with any prior systemic therapy for the treatment of active multiple myeloma. o Prior treatment of hypercalcemia or spinal cord compression with corticosteroids does not disqualify the patient (the dose should not exceed the equivalent of 320 mg of dexamethasone in a 2 week period). o Bisphosphonates are permitted. Prior Therapy for smoldering myeloma is permitted.
3. Patients treated with local radiotherapy with or without concomitant exposure to steroids, for pain control or management of cord/nerve root compression, are eligible. One week must have lapsed since last date of radiotherapy, which is recommended to be a limited field and from start of protocol therapy. . Patients who require concurrent radiotherapy should have entry to the protocol deferred until the radiotherapy is completed and one week have passed since the last date of therapy and from start of protocol therapy. .
4. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
5. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10-14 days prior to therapy and repeated again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
6. Age > / = 18 years at the time of signing Informed Consent.
7. Patients must meet the following laboratory criteria: absolute neutrophil count (ANC) >/= 1.5 x 10^9/L (growth factors not permitted to make eligible) , Hemoglobin >/= 9 g/dl (transfusion permitted) , Platelets >/= 100 x 10^9/L , Aspartate transaminase (AST) and Alanine transaminase (ALT) </= 2.5 x upper limits of normal (ULN) , Serum bilirubin </= 1.5 x ULN
8. Baseline Multi Gated Acquisition Scan (MUGA) or echocardiogram (ECHO) must demonstrate LVEF >/= 50%
9. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of </= 2
11. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

1. Patient has >/=Grade 2 peripheral neuropathy on clinical examination within 28 days of signing consent.
2. Renal insufficiency Creatinine > 2.5 mg/dl
3. Myocardial infarction within 6 months prior to signing consent or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any Electrocardiograph (ECG) abnormality at screening has to be documented by the investigator as not medically relevant.
4. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment.
5. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following: History or presence of sustained ventricular tachyarrhythmia; Any history of ventricular fibrillation or torsade de pointes; Bradycardia defined as HR< 50 bpm. Patients with pacemakers are eligible if heart rate (HR) >/= 50 bpm. Screening ECG with a QTcF > 450 msec, Right bundle branch block + left anterior hemiblock (bifascicular block) , Patients with myocardial infarction or unstable angina </= 6 months prior to starting study drug , Other clinically significant heart disease (e.g., congestive heart failure (CHF) New York Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
6. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat
7. Patients with diarrhea > Common Terminology Criteria for Adverse Events (CTCAE version 4) grade 2 at the time of signing consent
8. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
9. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
10. Female subject is pregnant or breast-feeding.
11. Hypersensitivity to acyclovir or similar anti-viral drug
12. Hypersensitivity to boron or mannitol, or compounds containing these components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-02-18 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Panobinostat with Bortezomib, Lenalidomide, and Dexamethasone | First 21 days of study drug administration (continuous dosing)
  Maximum tolerated dose (MTD) defined as highest dose level in which 6 participants have less than 2 instances of dose limiting toxicities (DLT). Toxicities graded in severity according to guidelines outlined in NCI-CTCAE version 4.0. Hematologic and non-hematologic DLTs defined differently, and will be based on experiences that occur during the first cycle of study drug administration.

SECONDARY OUTCOMES:
Overall Response Rate | After 8, 28 day cycles
  Response assessed according to the recently published International Uniform Response Criteria for multiple myeloma established by the International Myeloma Working Group (IMWG; Durie et al 2006).

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet E. Manasanch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Manasanch EE, Shah JJ, Lee HC, Weber DM, Thomas SK, Amini B, Feng L, Berkova Z, Hildebrandt M, Orlowski RZ. Bortezomib, lenalidomide, and dexamethasone with panobinostat for front-line treatment of patients with multiple myeloma who are eligible for transplantation: a phase 1 trial. Lancet Haematol. 2018 Dec;5(12):e628-e640. doi: 10.1016/S2352-3026(18)30174-1. PMID 30501870
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org